CLINICAL TRIAL: NCT06623773
Title: Prospective Non-Interventional Study on Structum® in Adult Patients With Osteoarthritis
Brief Title: Study on Structum® in Adult Patients With Osteoarthritis (TRUST)
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS13559
Record Dates: First submitted 2024-03-15; First posted 2024-10-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Chondroitin Sulfates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chondroitin sulfate — Chondroitin sulfate (CS) is a natural biomacromolecule belonging to the class of glycosaminoglycans and is an unbranched complex polysaccharide consisting of a repeating disaccharide structure of glucuronic acid and N-acetyl-D-glucosamine [18]. It is a major component of the extracellular matrix (ECM), where it constitutes an essential component of proteoglycans. Oral bioavailability of CS has been demonstrated [19], and its use for the treatment of OA has been established in animal models [20], as well as in clinical trials [21, 22]. CS, is available as a pharmaceutical grade drug (Structum®), meaning that the product is manufactured under Good Manufacturing Practices (GMP) conditions, and is in excess of 99% purity with no binders, fillers, excipients, dyes, or unknown substances. According to the Instructions for Use (IFU), the recommended posology for Structum® is 500 mg twice daily.
  Other Names: Structum

SUMMARY:
Chondroitin sulfate (CS) is a SYSADOA and a natural biomacromolecule belonging to the class of glycosaminoglycans. CS is a major component of the extracellular matrix (ECM), where it constitutes an essential component of proteoglycans.

To this date, no real-world studies have been conducted to precisely describe the burden associated with OA among patients treated with CS.Therefore, an observational, descriptive, prospective, national study will be conducted to describe the burden associated with OA and the quality of life of patients treated with Structum® in Poland.

DETAILED DESCRIPTION:
This is an observational, descriptive, national, multicentric, prospective, longitudinal study, which will be conducted over a 6-month follow-up period for each patient. The study will not provide or recommend any specific treatment or procedures.

All patients affected by OA in the knee, for whom Structum® is prescribed in a participating center, will be screened in a consecutive manner for eligibility. The study will focus exclusively on patients with OA in the knee as this is the joint most frequently affected and most easily assessed for OA patients.

Two additional data collections can be anticipated for these patients as part of their standard of care follow-up visits, which will usually occur around 3 and 6 months after the initial study visit.The patient enrolment period is expected to be 6 months, with a total study duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 50 to 80 years at inclusion
* of knee OA (either a patient newly diagnosed [at inclusion] or with history of knee OA) based on at least the following items 1 and/or 2:

  1. knee pain lasting for at least 3 months;
  2. patient in the active phase of knee OA disease (knee pain score ≥ 40mm at inclusion on the Visual Analog Scale [VAS] 0-100 mm);
  3. knee radiographs showing knee joint narrowing and/or osteophytes.
* Patients who have been prescribed, for the first time or not, Structum®.
* If patient is taking any NSAIDs or other analgesics, patient could be on stable dose at least one week before inclusion to the study.
* Patients able to visit the clinic and attend follow-up visits.
* Patients having signed an informed consent form, according to local regulations.

Exclusion Criteria:

* Patients with any ongoing chondroitin sulfate treatment at inclusion or during the last 3 months.
* plasma (in the last 3 months). No glucocorticoids administration in the last 3 months before inclusion. That does not include NSAIDS, paracetamol and other analgesic medications (e.g. tramadol).
* Patients with an artificial knee joint, including unilateral.
* Patients scheduled to undergo knee replacement surgery in the next 6 months.
* Patients with a severe general condition that prevents them from being included in the study as assessed by the investigator.
* Patients participating in interventional trials on investigational drugs at the time of inclusion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged 50 to 80 years with a confirmed diagnosis of knee osteoarthritis and a new prescription for Structum®, as treated by participating centers in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
describe the baseline clinical profile and baseline OA symptom severity (pain, stiffness and function) as assessed by the (WOMAC) questionnaire, for patients with knee OA and treated with Structum®. | baseline
  description at enrollment of Demographics and clinical characteristics of patients with knee OA- description of treatment history- description of knee OA symptm severity per the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  The total WOMAC score range is from 0-2400, with higher scores indicating worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Secondary Womac outcomes at 3-months | from baseline to 3 months after baseline
  Mean global score of symptoms severity of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  The total WOMAC score range is from 0-2400, with higher scores indicating worse pain, stiffness, and functional limitations.
Secondary Womac outcomes at 3-months | from baseline to 3 months after baseline
  Mean score of each dimension of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  For each dimension, the values scored on each item will be summed to give a dimension score, with pain ranging from 0-500, stiffness 0-200, and physical function 0-1700.
Secondary Womac outcomes at 3-months | from baseline to 3 months after baseline
  Mean difference in symptoms severity score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
Secondary Womac outcomes at 6-months | from baseline to 6 months after baseline
  Mean difference in symptoms severity score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  The total WOMAC score range is from 0-2400, with higher scores indicating worse pain, stiffness, and functional limitations.
Secondary Womac outcomes at 6-months | from baseline to 6 months after baseline
  Mean score of each dimension of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  For each dimension, the values scored on each item will be summed to give a dimension score, with pain ranging from 0-500, stiffness 0-200, and physical function 0-1700.
Secondary Womac outcomes at 6-months | from baseline to 6 months after baseline
  Mean global score of symptom severity of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC )Questionnaire.
  The total WOMAC score range is from 0-2400, with higher scores indicating worse pain, stiffness, and functional limitations.
Bone's outcome at baseline | baseline
  Mean global score of the OA burden of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
Bone's outcome at baseline | baseline
  Mean score of each dimension of the Burden Osteoarthritis New'Scale (BONe'S) Each question (19 questions) of each dimension is evaluated from to 5.
Bone's outcome at 3 months | from baseline to 3 months after baseline
  Mean global score of the OA burden of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
Bone's outcome at 6 months | from baseline to 6months after baseline
  Mean global score of the OA burden of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
Bone's outcome at 3 months | from baseline to 3 months after baseline
  Mean score of each dimension of the Burden Osteoarthritis New'Scale (BONe'S) Each question (19 questions) of each dimension is evaluated from to 5.
Bone's outcome at 6 months | from baseline to 6 months after baseline
  Mean score of each dimension of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
Bone's outcome at 3 months | from baseline to 3 months after baseline
  Mean difference in OA burden scores at 3 months of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
Bone's outcome at 6 months | from baseline to 6 months after baseline
  Mean difference in OA burden scores at 6 months of the Burden Osteoarthritis New'Scale (BONe'S) The total score range is 0-100 scale. Higher scores represent a heavier burden
SF12 outcome at baseline | baseline
  mean global score of general health of the Short Form Questionnaire (SF12) Scores range from 0 to 100, with higher scores indicating a better physical and mental health functioning.
SF12 outcome at 3 months | from baseline to 3 months after baseline
  mean global score of general health of the Short Form Questionnaire (SF12) Scores range from 0 to 100, with higher scores indicating a better physical and mental health functioning.
SF12 outcome at 6 months | from baseline to 6 months after baseline
  mean global score of general health of the Short Form Questionnaire (SF12) Scores range from 0 to 100, with higher scores indicating a better physical and mental health functioning.
SF12 outcome at baseline | baseline
  mean score of physical and mental dimension of the Short Form Questionnaire (SF12) A special scoring program, accessible via the license purchase of the questionnaire, will be used to analyze this questionnaire by giving a ponderation to each item to result in two different dimension scores.
SF12 outcome at 3 months | from baseline to 3 months after baseline
  mean score of physical and mental dimension of the Short Form Questionnaire (SF12) A special scoring program, accessible via the license purchase of the questionnaire, will be used to analyze this questionnaire by giving a ponderation to each item to result in two different dimension scores
SF12 outcome at baseline at 6 months | from baseline to 6 months
  mean score of physical and mental dimension of the Short Form Questionnaire (SF12) A special scoring program, accessible via the license purchase of the questionnaire, will be used to analyze this questionnaire by giving a ponderation to each item to result in two different dimension scores
Persitence outcomes at 3 months | from baseline to 3 months after baseline
  proportion of patients with ongoing Structum® at 3 months
Persitence outcomes at 6 months | from baseline to 6 months after baseline
  proportion of patients with ongoing Structum® at 6 months
Personal global assessment, after first dose of Structum®, at 3 months | from baseline to 3 months after baseline
  Proportion of patients with a positive assessment of Structum®, as assessed by Structum® treatment satisfaction questionnaire
Personal global assessment, after first dose of Structum®, at 6 months | from baseline to 6 months after baseline
  Proportion of patients with a positive assessment of Structum®, as assessed by Structum® treatment satisfaction questionnaire

OTHER OUTCOMES:
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the SF-12 questionnaire at inclusion. | baseline
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the SF-12 questionnaire at 3 months | from baseline to 3 months after baseline
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the SF-12 questionnaire at 6 months | from baseline to 6 months after baseline
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the WOMAC questionnaire at inclusion | baseline
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the WOMAC questionnaire at 3 months | from baseline to 3 months after baseline
Spearman correlation coefficient and P value for the correlation between the BONe'S questionnaire and the WOMAC questionnaire at 6 months. | from baseline to 6 months after baseline
Variables of interest for the assessment of this exploratory outcome will originate from the BONe'S, SF-12 and WOMAC questionnaires | from baseline to 6 months after baseline
  Calculation of the Spearman correlation coefficient at inclusion, 3, and 6 months for the correlation between
  * the BONe'S questionnaire (the independence + interaction & recreation + hygiene & beauty scores) and the SF-12 questionnaire (physical component summary dimension).
  * the BONe'S questionnaire (psychological score) and the SF-12 questionnaire (mental component summary dimension)
  * the global score of the BONe'S questionnaire and the total WOMAC score.
Proportion of patients with changes in the prescription of NSAIDs and other analgesics 6 months before inclusion, at inclusion | baseline
  Description of the proportion of patients with a change in their prescription of NSAIDs and other analgesics 6 months before inclusion, at inclusion, and at 3 and 6 months, with a change being defined as any change of the daily dose of NSAIDs (calculated from the frequency of intake and the dose of each intake)
  * Increased
  * Stable
  * Decreased
Proportion of patients with changes in the prescription of NSAIDs and other analgesics 6 months before inclusion, at 3 months | from baseline to 3 months after baseline
Proportion of patients with changes in the prescription of NSAIDs and other analgesics 6 months before inclusion, at 6 months | from baseline to 6 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: PIOTR WILAND, Principal Investigator — Medical University of WROCLAW
Locations (15):
- Poland (15):
  - Maciej Dołżyński, Bialystok
  - Piotr Ligocki, Bydgoszcz
  - Elżbieta Pietrus- Dunaszewska, Katowice
  - Bartlomiej Szpyra, Krakow
  - Alina Wołkowicz Mruk, Krakow
  - Andrzej Majer, Kujakowice Gorn
  - Agnieska WIAK, Lubartów
  - Wojciech Larczyński, Nowy Dwór Gdański
  - Sławomir Panek, Olesno
  - Marcin Milchert, Szczecin
  - Wojciech Roczniak, Ustrzyki Dolne
  - Zdzisław Derleta, Warsaw
  - Michał Straburzyński, Zielona Góra
  - Mariusz Borowiecki, Zielona Góra
  - Viktor Kostiuk, Żagań

IPD SHARING:
Plan to Share IPD: No
Data will be collected and retained in a pseudonymized format, with no directly identifying values that might link the data to the corresponding participant to the study.
  The Investigator must ensure that the patient's confidentiality is maintained. It is required that the Investigator and institution permit authorized representatives of the Sponsor, of the regulatory agency(s), and the institutional ECs direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study.